CLINICAL TRIAL: NCT06330532
Title: Impact of Preoperative Frailty and Cognitive Impairment on Postoperative Outcomes in Elderly Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-1526
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients categorized as having no frailty on the frailty item, assessed by four domains: cognitive, emotional, physical, and nutritional.
- Patients exhibiting the early signs that may lead to frailty, assessed in four domains: cognitive, emotional, physical, and nutritional.
- Patients categorized as having frailty on the frailty item, assessed by four domains: cognitive, emotional, physical, and nutritional.

SUMMARY:
This is a retrospective study of patients aged 65 years and older who underwent cardiac and aortic surgery between March 5, 2021 and October 12, 2022 in the operating room of Severance Cardiovascular Hospital to determine the impact of physical frailty as well as nutritional status, emotional dysregulation, and cognitive dysfunction on postoperative outcomes. Physical frailty will be determined by the Clinical Frailty Scale, handgrip strength, and nutritional status, cognitive dysfunction will be determined by the K-MMSE and K-MoCA administered at the preoperative interview, and emotional dysregulation will be determined using the SGDS-K. These were measured during the pre-anesthesia evaluation and only results from patients who agreed to be tested will be used. Nutritional status will be analyzed based on blood test values measured within one month of surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65-year-old patients undergoing surgery for heart and aortic disease, who completed physical (Clinical Frailty scale, Handgrip strength), cognitive(K-MoCA, K-MMSE), and emotional (SGDS-K) functioning tests at the preoperative interview

Exclusion Criteria:

* Failed to complete two or more of assessments shown above

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients age 65 and older undergoing heart and aortic surgery
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
postoperative all cause mortality | within 1 year
  This study evaluates all-cause mortality within 1 year after surgery
major composite morbidity | within 30days after surgery for major composite morbidity

SECONDARY OUTCOMES:
the number of days not in hospital | 90 days
  DAOH is the number of days not in hospital over a defined postoperative period
The number of participants who die | 30 days after surgery
  patients who die

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea